CLINICAL TRIAL: NCT02202967
Title: Misoprostol for the Healing of Small Bowel Ulceration in Patients With Obscure Blood Loss While Taking Low-dose Aspirin or Nonsteroidal Antiinflammatory Drugs [MASTERS Trial]
Brief Title: Misoprostol for Small Bowel Ulcers and Obscure Bleeding Due to Aspirin or Nonsteroidal Antiinflammatory Drugs
Acronym: MASTERS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN09CA403; 2013-003187-31 (EudraCT Number)
Record Dates: First submitted 2014-07-26; First posted 2014-07-29 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Chronic Arthritis; Ischemic Heart Disease; Atrial Fibrillation; Anemia; Bleeding
Keywords: Aspirin; Intestinal bleeding; Misoprostol; NSAIDs; Small intestine; Video capsule endoscopy
MeSH Terms: conditions — Myocardial Ischemia; Atrial Fibrillation; Anemia; Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): Misoprostol
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Misoprostol oral tablets/ capsules contain 200 mcg of Misoprostol, a synthetic prostaglandin E1 analog
  Other Names: Cytotec (R)
  Arms: Misoprostol
Drug: Placebo — Placebo contains lactose granules
  Other Names: Dummy drug
  Arms: Placebo

SUMMARY:
Anti-inflammatory tablets (non-steroidal anti-inflammatory drugs) continue to be used commonly worldwide to relieve pain caused by arthritis. Likewise, aspirin is used by many patients in order to prevent blood clots. Despite their desired benefits, these medicines can cause internal bleeding from the digestive system. The source of this bleeding can be obvious (overt), or obscure and thought to come from the small intestine. Obscure bleeding can show as anemia due to lack of iron in the blood. Small intestine ulcers are now easily diagnosed using an endoscope the size of a big pill (video capsule endoscopy). Small bowel ulcers are not related to stomach acid and therefore do not heal using remedies usually taken to stop acid formation. A different drug, misoprostol, consists of a chemical (prostaglandin) that is usually lacking in patients using aspirin or anti-inflammatory drugs. Misoprostol is licenced to heal stomach and duodenal ulcers in patients using these drugs. Our hypothesis is that misoprostol might be effective in healing small bowel ulcers as suggested by pilot studies; however, such works only included small numbers of patients, did not include control groups and both patients and investigators knew the nature of the tablets used. To test this hypothesis, we propose to compare misoprostol to a dummy tablet. The numbers of subjects to be studied have been calculated using established statistical methods

DETAILED DESCRIPTION:
METHODOLOGY:

* Upper gastrointestinal endoscopy and colonoscopy on patients with obscure bleeding and/ or iron deficiency anemia.
* Video capsule endoscopy on those fulfilling the inclusion criteria
* Randomization to Misoprostol 200 micrograms or placebo, 4 times each day given for 8 weeks to aspirin/ NSAID users with erosive small bowel lesions.
* Video capsule endoscopy at 8 weeks to check healing of small bowel lesions.
* Full blood count at baseline and monthly intervals (0, 4, and 8 weeks)

ELIGIBILITY:
INCLUSION CRITERIA:

Obscure occult gastrointestinal bleeding: presence of one or more of the following:

* Positive fecal occult blood test within last 3 months
* Iron deficiency anemia (ferritin <100 ug/l, hemoglobin [Hb] 7-12 g/dl [female] or 7-13 g/dl [male])
* Drop in haemoglobin, > 2gm/dl from baseline, in the absence of potential or actively bleeding lesion detectable on upper endoscopy or colonoscopy.

Normal/ absence of potentially bleeding lesions on full upper endoscopy and colonoscopy.

Taking low-dose aspirin (75-325m/ day) and/ or NSAIDs

MAIN EXCLUSION CRITERIA:

* Incomplete upper endoscopy or colonoscopy
* Systemic disease that is unstable at the time of randomisation (unstable vital signs; ongoing non-gastrointestinal investigations; frequent modifications to treatment)
* Intake of certain drugs: high-dose steroids (>7.5-mg prednisolone/ day), cytotoxic drugs, or warfarin.
* Upper gastrointestinal lesions: oesophageal varices; oesophageal stricture; oesophageal or gastric neoplasms; pyloric stenosis; peptic ulcers; vascular malformations.
* Colonic disorders: neoplasms or adenomatous polyps; inflammatory bowel disease; vascular malformations; actively bleeding diverticular disease
* Women planning pregnancy, pregnant or women of child-bearing potential not using two contraceptive methods, one of which must be highly effective [implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner]
* Hypotension: systolic blood pressure <100-mm Hg.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Full healing of small bowel mucosal ulcers or erosions in response to misoprostol in users of aspirin or NSAIDs. | 8 weeks
  Ulcers or smaller lesions (erosions) should totally disappear by the end of the study

SECONDARY OUTCOMES:
Change in the numbers of mucosal ulcers and erosions | 8 weeks
  Any increase or decrease in the numbers of ulcers and erosions will be measured at the end of the study

OTHER OUTCOMES:
Change in blood haemoglobin level | 8 weeks
  Any rise or drop in the haemoglobin level will be measured at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Travers, PhD, Study Director — NHS Greater Glasgow & Clyde, Scotland
Locations (1):
- University Hospital Crosshouse, Kilmarnock, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taha AS, McCloskey C, McSkimming P, McConnachie A. Misoprostol for small bowel ulcers in patients with obscure bleeding taking aspirin and non-steroidal anti-inflammatory drugs (MASTERS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Jul;3(7):469-476. doi: 10.1016/S2468-1253(18)30119-5. Epub 2018 May 10. PMID 29754836
- See also: Taha AS et al. MASTERS Trial.Lancet Gastroenterol Hepatol 2018;3:469-76 — http://dx.doi.org/10.1016/S2468-1253(18)30119-5